CLINICAL TRIAL: NCT00832871
Title: INST 0817: Compassionate Use of Mifepristone
Brief Title: Compassionate Use of Mifepristone in Brain/Nervous System and Other Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual; 4 patients enrolled between 2008-2015
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: The Feminist Majority Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: INST 0817; NCI-2011-02682 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Cancer
Keywords: Mifepristone; RU-486; Compassionate Use; Antiprogesterone
MeSH Terms: conditions — Neoplasms | interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mifepristone (Experimental): 200 mg RU-486 (Mifepristone) daily
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 200 mg will be administered orally
  Other Names: RU-486; Mifeprex

SUMMARY:
The purpose of this study is to see if mifepristone prevents worsening of your cancer. Mifepristone is an antiprogesterone agent, a drug which blocks female hormones, that is commonly used for the termination of pregnancies. It has not been approved by the Food and Drug Administration for use in the treatment of cancer. It is unlicensed in the United States for your condition. However, previous work has indicated that mifepristone may be useful due to how it works. It is being made available for use in the United States for compassionate use through the Feminist Majority Foundation.

DETAILED DESCRIPTION:
This is a compassionate use of mifepristone treatment for patients with conditions that could respond to an antiprogesterone agent, including:

* Meningioma.
* Breast cancer
* Colon Cancer
* Endometrial Stromal Sarcoma
* Bilateral Chronic Central Serous Retinopathy
* Cushing's Syndrome
* Metastatic Adrenocortical Cancer
* Ovarian Cancer
* Other conditions as determined by the attending physicians

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older.
* Patients must sign an informed consent.
* Patients should be in such a health condition in the opinion of the attending physician that with the administration of mifepristone benefits may outweigh risks.

Exclusion Criteria:

* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Chyi Lee, M.D., Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- Universtiy of New Mexico - Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mifepristone
Number analyzed (Participants) | 4
Age, Continuous [Median (Full Range); unit: years] | 45 [25 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Duration of Response
Description: The time from the date of response (not the beginning of treatment unless there is stable disease) to disease progression. Response and progression are evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.0). Target lesions are assessed by computerized tomography (CT) or magnetic resonance imaging (MRI): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient decrease in the sum of the longest diameter of target lesions to qualify for PR nor sufficient increase in the sum of the longest diameter of target lesions to qualify for Progressive Disease; Progressive Disease (PD), 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 5 years
Population: Only one patient achieved stable disease. This patient's duration of response could therefore be reported. The other three patients progressed on treatment.
Measure: Median (Full Range); unit: days
Arm/Group | Mifepristone
Number analyzed (Participants) | 1
days | 44 [44 to 44]

2. Secondary Outcome: Toxicity Associated With Adrenal Insufficiency
Description: Toxicity will be evaluated per National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE), version 3.0. Frequency and severity of adverse events will be tabulated using counts the following events of interest, which are related to possible adrenal insufficiency: nausea, vomiting, lethargy, dizziness, fatigue, anorexia, and skin rash. Any grade of these events that are self-reported by patients as well as events identified by physician assessment (e.g. physical exam) will be included.
Time Frame: Up to 8 weeks after the end of study treatment or until any adverse events are resolved (whichever is longest)
Population: All patients received at least one dose of study medication and are included in this analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 4
percentage of participants
  Nausea | 0
  Vomiting | 0
  Lethargy | 0
  Dizziness | 0
  Fatigue | 0
  Anorexia | 0
  Skin Rash | 0

3. Other Pre Specified Outcome: Overall Survival
Description: The time from patient entry into the protocol to death by any cause.
Time Frame: 5 years
Measure: Median (Standard Deviation); unit: Months
Arm/Group | Mifepristone
Number analyzed (Participants) | 4
Months | 24.2 (28.5)

ADVERSE EVENTS:
Arm/Group | Mifepristone
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=4)
Edema: limb (Blood and lymphatic system disorders) | 1 (1)
Edema: trunk (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Watery eye (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This is a compassionate use protocol. No statistical analysis was specified in the protocol; it states that only descriptive data will be collected. Data from only 4 patients should not be considered reliable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No